CLINICAL TRIAL: NCT03110588
Title: Phase I Trial of Prednisone, Abiraterone, Cabazitaxel and Enzalutamide (PACE) for Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Phase I Trial of PACE for Metastatic Prostate Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Astellas Pharma Inc (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F161215003 (UAB 1663)
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Prostate Cancer
Keywords: metastatic prostate cancer; castration-resistant prostate cancer; PACE (Prednisone, Abiraterone, Cabazitaxel, and Enzalutamide)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel

STUDY DESIGN:
Intervention Model Description: The first cohort will administer the following to three patients: prednisone 5 mg orally twice daily, abiraterone 1000 mg orally once daily, enzalutamide 160 mg orally once daily, and cabazitaxel intravenous infusion at 15 mg/m2 every 3 weeks. If there are no dose limiting toxicities, the cabazitaxel will be escalated to 20 mg/m2 in a second cohort. The other three drugs will remain at the same dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PACE with Cabazitaxel @ 15 mg/m2 (Experimental): The drugs to be administered are: prednisone 5 mg orally twice daily, abiraterone 1000 mg orally once daily, enzalutamide 160 mg orally once daily, and cabazitaxel intravenous infusion at 15 mg/m2 every 3 weeks.
  Interventions: Drug: PACE with Cabazitaxel (15 mg/m2)
- PACE with Cabazitaxel @ 20 mg/m2 (Experimental): The drugs to be administered are: prednisone 5 mg orally twice daily, abiraterone 1000 mg orally once daily, enzalutamide 160 mg orally once daily, and cabazitaxel intravenous infusion at 20 mg/m2 every 3 weeks.
  Interventions: Drug: PACE with Cabazitaxel (20 mg/m2)

INTERVENTIONS:
Drug: PACE with Cabazitaxel (15 mg/m2) — Prednisone, Abiraterone, and Enzalutamide are administered orally; Cabazitaxel is be administered intravenously @ 15 mg/m2.
  Arms: PACE with Cabazitaxel @ 15 mg/m2
Drug: PACE with Cabazitaxel (20 mg/m2) — Prednisone, Abiraterone, and Enzalutamide are administered orally; Cabazitaxel is be administered intravenously @ 20 mg/m2.
  Arms: PACE with Cabazitaxel @ 20 mg/m2

SUMMARY:
This trial is being conducted to determine the feasibility and recommended dose of the combination of four drugs (prednisone, abiraterone, cabazitaxel and enzalutamide (PACE) as first-line therapy for metastatic castration-resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
Multiple agents have been shown to improve survival in patients with mCRPC by up to five months. The combination of prednisone, abiraterone, cabazitaxel and enzalutamide may be anticipated to be feasible therapy with minimal or no adverse drug interactions. This is a phase I trial to study the feasibility of the proposed therapy.

Patients will undergo a combination of oral daily drug intake at varying doses over a period of three weeks. Monitoring including blood collection for laboratory testing will be done on Day 1 of each three-week cycle with additional monitoring during the first cycle. Imaging and correlative studies will be done every 12 weeks. Therapy will continue until disease progression or severe toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Histologically proven adenocarcinoma of the prostate with metastatic disease.
3. Progressive disease following androgen deprivation therapy; Prostate Specific Antigen (PSA) progression defined as baseline increase followed by any PSA increase greater than or equal to 1 week apart.
4. Most recent PSA ≥2 ng/ml
5. Testosterone < 50 ng/dL
6. Anti-androgen withdrawal of first generation AR inhibitors (bicalutamide, nilutamide) is required for 6 weeks if previous duration of stability on them was ≥3 months.
7. ECOG performance status 0-1.
8. Adequate organ function as defined below:

   ANC 1,500/µl; Hemoglobin 10 g/dL; Platelet count 100,000/µL; Creatinine clearance ≥45 ml/min; Potassium >3.5 mmol/L (or within institutional normal range) Bilirubin ≤ ULN (unless documented Gilbert's disease); SGOT (AST) 1.5 x ULN; SGPT (ALT) 1.5 x ULN
9. Subject agrees to use a double barrier method of contraception during the course of study therapy and for at least 3 months after completion of therapy. A double barrier method involves the use of a condom in combination one of the following: sponge, diaphragm, cervical ring with spermicidal gel or foam. Subjects who have had a vasectomy ≥6 months prior to trial therapy and those with female sexual partners who are 55 years old and post-menopausal for 2 years or sterile (by tubectomy, hysterectomy, bilateral oophorectomy) need to agree to use at least a condom.
10. Ability to sign a written informed consent form.
11. Subject is willing to stop herbal supplements.

Exclusion Criteria:

1. Prior docetaxel for castration-resistant disease (prior docetaxel for castration-sensitive disease is allowed but not required).
2. Prior enzalutamide, abiraterone, cabazitaxel.
3. History of severe hypersensitivity reaction (≥grade 3) to docetaxel.
4. History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs.
5. Concomitant vaccination with yellow fever vaccine.
6. Prior investigational androgen synthesis or androgen receptor antagonists.
7. Prior hypersensitivity reaction to capsule components of enzalutamide including labrasol, butylated hydroxyanisole and butylated hydroxytoluene
8. Other non-chemotherapeutic investigational agents within 14 days (prior chemotherapy needs a ≥4 week washout).
9. Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments).
10. Prior isotope therapy with Strontium-89, Samarium or radium-223.
11. Patients with a history of central nervous system metastases (brain, meninges, spinal cord).
12. Imminent risk of pathologic fracture or cord compression.
13. History of seizures, underlying brain injury with loss of consciousness, transient ischemic attack within 12 months, cerebrovascular accident, and brain arteriovenous malformations.
14. Uncontrolled severe intercurrent illness or medical conditions including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III and IV heart failure), unstable angina pectoris, uncontrolled diabetes mellitus, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or concurrent medications that alter cardiac conduction.
15. Patients with a "currently active" second malignancy other than non- melanoma skin or superficial urothelial cancers are not eligible. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are now considered without evidence of disease for 3 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The patient must have a cancerous prostate.
Enrollment: 0 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of PACE as first-line therapy | Baseline up to 2 years
  The maximum tolerated dose is when 6 patients are treated at a dose level with less than two patients demonstrating dose limiting toxicities. Dose limiting toxicities are defined as any grade greater than or equal to grade 3 non-hematologic toxicity (except greater than or equal to grade 2 neurotoxicity), or greater than or equal to grade 4 neutropenia or thrombocytopenia lasting longer than or equal to 7 days. Toxicities will be assessed according to the NCI Common Terminology Criteria for Adverse Events version 4.03.

SECONDARY OUTCOMES:
Prostate specific antigen (PSA) | Baseline up to 2 years
  PSA with a greater than or equal to 30% result within 12 weeks from baseline or the previous result and maximum declines at any time during the study progression. PSA will be tested at least every 3 weeks.
Radiographic progression-free survival with PACE | Baseline up to 2 years
  Radiographic examination is performed every 12 weeks to determine if there is disease progression.
Progression-free survival with PACE | Baseline up to 2 years
  Progression-free survival is defined as the duration of time from start of treatment to time of progression or death, whichever comes first.
Objective response rate of measurable disease | Baseline up to 2 years
  Response will be evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria. Target lesions should be selected based on size (lesions with the longest diameter) and their suitability for accurate repeated measurements. A sum of the longest diameter (LD) for all target lesions will be calculated and reported as the baseline sum LD, which will be used to characterize the objective tumor response.
Pain response | Baseline up to 2 years
  The Patient Pain Index (0-5 scale) is used to measure pain per cycle. A decline of greater than or equal to 2 is defined as pain response.

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor N Saleh, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No